CLINICAL TRIAL: NCT01691963
Title: Epiglottic Downfolding During Endotracheal Intubation - An Alternative Technique to Improve Glottic Exposure and Facilitate Intubation?
Brief Title: Epiglottic Downfolding During Endotracheal Intubation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Main investigators (Pieters/van Zundert) changed institutions. Therefore, they were not able to start the study and decided to withdraw the study for now.
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Barbe Pieters, Principal investigator, Catharina Ziekenhuis Eindhoven
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: M12-1233; NL40875.060.12 (Other: Medisch Ethische Commissie Catharina Ziekenhuis Eindhoven)
Record Dates: First submitted 2012-09-19; First posted 2012-09-25 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Intubation Complication; Injury of Epiglottis
Keywords: Epiglottis; Intubation; Laryngoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): In the control group, anaesthesia will be induced in the same way as mentioned above for the intervention group. Also in this group, intubation will be achieved using a C-MAC® videolaryngoscope (Karl Storz, Tuttlingen, Germany) with a size 3 Macintosh blade.
  The best possible view of the glottic inlet will be scored with the blade tip positioned in the vallecula. The glottic view will be scored in this position using the Cormack and Lehane classification system. If correct laryngoscope positioning cannot be achieved with a size 3 blade, a size 4 blade will be used. Hereafter, the patient's trachea will be intubated once the optimal view of the larynx had been obtained. Intubation attempts will be scored in the same way as mentioned above for the intervention group.
- Epiglottic downfolding (Experimental): Endotracheal intubation will be achieved using a C-MAC® videolaryngoscope (Karl Storz, Tuttlingen, Germany) with a size 3 Macintosh blade.
  The best possible view of the glottic inlet will be scored with the blade tip positioned in the vallecula.
  Next, the view of the glottic inlet will be scored with the blade advanced further into the vallecula, until the epiglottis flips infero-posteriorly and becomes downfolded into the trachea.
  The glottic view will be scored in both positions using the Cormack and Lehane classification system.
  After successful intubation, the blade will slowly be withdrawn into the vallecula to elevate the epiglottis back to its normal position.
  Interventions: Device: C-MAC® videolaryngoscope (Karl Storz, Tuttlingen, Germany)

INTERVENTIONS:
Device: C-MAC® videolaryngoscope (Karl Storz, Tuttlingen, Germany) — Endotracheal intubation will be achieved using a C-MAC® videolaryngoscope (Karl Storz, Tuttlingen, Germany) with a size 3 Macintosh blade.
  The best possible view of the glottic inlet will be scored with the blade tip positioned in the vallecula.
  Next, the view of the glottic inlet will be scored with the blade advanced further into the vallecula, until the epiglottis flips infero-posteriorly and becomes downfolded into the trachea.
  The glottic view will be scored in both positions using the Cormack and Lehane classification system.
  After successful intubation, the blade will slowly be withdrawn into the vallecula to elevate the epiglottis back to its normal position.
  Other Names: Epiglottic downfolding during endotracheal intubation
  Arms: Epiglottic downfolding

SUMMARY:
Usually videolaryngoscopy using a videolaryngoscope with a classic Macintosh design is performed with the blade in the vallecula and the epiglottis elevated from the vocal cords indirectly, as in direct laryngoscopy. However, during an audit of videolaryngoscopic practice we noticed that, in obtaining the best view, clinicians frequently and inadvertently advanced the blade into the vallecula to get a better view, such that the epiglottis was downfolded and elevated directly from the vocal cords. However, a better view does not necessarily lead to higher intubation success.

In this randomized, controlled trial, we want to determine the efficacy of videolaryngoscope-guided tracheal intubation using an alternative position for the blade in patients with normal airways.

DETAILED DESCRIPTION:
Anaesthesia will be induced in the conventional matter. For patients randomized to the intervention group, when the anaesthesiologist considers the depth of anaesthesia to be sufficient, a C-MAC® videolaryngoscope (Karl Storz, Tuttlingen, Germany), will be placed into the patients mouth. The best possible view of the vocal cords will be obtained with the blade positioned normally in the vallecula anterior to the epiglottis. The epiglottis will be elevated from the vocal cords indirectly, identical with direct laryngoscopy. After this, the best possible view of the vocal cords will be obtained with the blade positioned alternatively in the vallecula posterior to the epiglottis, such that the epiglottis is downfolded and elevated directly from the vocal cords. Views will be scored in both positions using the Cormack and Lehane classification system. When correct laryngoscope positioning can't be achieved with a size 3 blade, a size 4 blade will be used.

For patients not randomized to the intervention group, anaesthesia will also be induced in the conventional matter. When the anaesthesiologist considers the depth of anaesthesia to be sufficient, a C-MAC® videolaryngoscope (Karl Storz, Tuttlingen, Germany), will be placed into the patients mouth. The best possible view of the vocal cords will be obtained with the blade positioned normally in the vallecula anterior to the epiglottis. The epiglottis will be elevated from the vocal cords indirectly, identical with direct laryngoscopy. The view will be scored in this position using the Cormack and Lehane classification system. After this, the patient will be intubated.

Patients will be interviewed 2 and 24 hours postoperatively about sore throat, dysphonia, dysphagia and coughing.

ELIGIBILITY:
Inclusion Criteria:

* Informed patient consent
* ASA I-III
* Age > 18 years
* Elective surgery, other than head and/or neck surgery
* Elective surgery, duration < 1 hour in supine position
* Pre-operative Mallampati I-II-III

Exclusion Criteria:

* No informed patient consent
* ASA IV
* Age < 18 years
* Preoperative complaints of sore throat, dysphagia, dysphonia and coughing
* Emergency surgery, surgery of head and/of neck
* Surgery during > 1 hour in other than supine position
* Locoregional anaesthesia
* Preoperative Mallampati IV
* Known difficult airway
* Bad dentition
* Dental crowns and/or fixed partial denture
* Risk of aspiration (fasted < 6 hours, gastroesophageal reflux)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
The Cormack and Lehane grade | Patients will be followed for the duration of induction of anaesthesia, an average of 10 minutes
  The Cormack and Lehane grade scored in both positions of the C-MAC® videolaryngoscope and consequent success of intubation

SECONDARY OUTCOMES:
Discomfort | Patients will be followed for 24 hours postoperatively
  Sore throat, dysphonia, dysphagia and coughing reported by patients 2 and 24 hours postoperatively
Use of adjuncts | Patients will be followed for the duration of induction of anaesthesia, an average of 10 minutes
  Frequency of use of a stylet, gum elastic bougie or BURP manoeuvre.

CONTACTS AND LOCATIONS:
Overall Officials: Barbe MA Pieters, MD, Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (1):
- Catharina Ziekenhuis Eindhoven, Eindhoven, Netherlands

REFERENCES:
- [Background] van Zundert A, van Zundert T, Brimacombe J. Downfolding of the epiglottis during intubation. Anesth Analg. 2010 Apr 1;110(4):1246-7. doi: 10.1213/ANE.0b013e3181ce716f. No abstract available. PMID 20357168
- [Background] Kaplan MB, Hagberg CA, Ward DS, Brambrink A, Chhibber AK, Heidegger T, Lozada L, Ovassapian A, Parsons D, Ramsay J, Wilhelm W, Zwissler B, Gerig HJ, Hofstetter C, Karan S, Kreisler N, Pousman RM, Thierbach A, Wrobel M, Berci G. Comparison of direct and video-assisted views of the larynx during routine intubation. J Clin Anesth. 2006 Aug;18(5):357-62. doi: 10.1016/j.jclinane.2006.01.002. PMID 16905081
- [Background] Merli G. Videolaryngoscopy: is it only a change of view? Minerva Anestesiol. 2010 Aug;76(8):569-71. Epub 2010 Apr 23. No abstract available. PMID 20661194